CLINICAL TRIAL: NCT02216344
Title: Controlled Acute Hypoxia Study Comparing Pulse Oximetry to Arterial Blood Samples Using the Abbreviated Sensor Line in Healthy Subjects With the USB Pulse Oximetry Monitor Interface Cable
Brief Title: Controlled Acute Hypoxia Study - Abbreviated Sensor Line
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0440
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Healthy; Hypoxia
Keywords: Patient safety monitors
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulse Oximeter (the device): The pulse oximetry devices were placed on subjects per the protocol. The subjects underwent gradual hypoxia and the output of the devices under test was compared to the SaO2 value as measured by a CO-Oximeter (the reference value), as outlined by ISO 80601, to ensure that the devices meet the specified performance claims.

SUMMARY:
The primary objective of the study is to validate the proposed claims for the OxiCable device, for pulse rate and saturation accuracy in a diverse subject population over a specified saturation range.

DETAILED DESCRIPTION:
The general procedure of invasive controlled hypoxia clinical studies is to directly compare test pulse oximeter measurements to saturation measurements made by a multi-wavelength CO-oximeter taken from arterial blood samples from healthy human subjects. Following arterial cannulation, hypoxia is induced by reducing the percent of inspired oxygen the subject breathes while simultaneous measurements are recorded from the test pulse oximeters and arterial blood samples at targeted levels of saturation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race
* 18-50 years old, inclusive
* Females: negative urine pregnancy test on the day of study participation (prior to exposure to hypoxia)
* Completed within the last year: physical exam by a licensed physician, physician assistant (PA), or advanced practice nurse; including a 12 lead ECG, a medical history, and blood test (complete blood count and sickle cell trait/disease screening)
* Meets specific demographic requirements for the monitoring device under study
* Willing and able to provide written informed consent
* Able to participate for the duration of the evaluation

Exclusion Criteria:

* Under 18 years or over 50 years of age
* Pregnant and/or lactating women
* Hypertension: on three consecutive readings, systolic pressure greater than 145 mm Hg or diastolic pressure greater than 90 mm Hg
* Premature ventricular contractions (PVCs) that are symptomatic or occur at a rate of more than four per minute
* History of seizures (except childhood febrile seizures) or epilepsy
* History of unexplained syncope
* Daily or more frequent use of anxiolytic drugs (benzodiazepines) for treatment of anxiety disorder
* Recent history of frequent migraine headaches: average of two or more per month over the last year
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test site needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* History of acute altitude sickness at or below moderate elevation (up to 5,000-10,000 feet) defined as three or more of the following symptoms: moderate to severe headache, general malaise, dizziness/lightheadedness, nausea/vomiting, fatigue/weakness, shortness of breath, nosebleed, persistent rapid pulse, or peripheral edema
* History of significant respiratory disease such as severe asthma or emphysema
* Sickle cell disease or trait
* Clinically significant abnormal finding on medical history, physical examination, clinical laboratory test or ECG. Clinical significance will be assessed by the principal investigator or study physician as designated.
* History of stroke, transient ischemic attack or carotid artery disease
* History of myocardial ischemia, angina, myocardial infarction, congestive heart failure or cardiomyopathy
* History of chronic renal impairment
* Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
* Unwillingness or inability to remove colored nail polish from test digit(s)
* Unwillingness or inability to give informed consent
* Prior or known allergies to: lidocaine (or similar pharmacological agents, e.g., Novocain) or heparin
* Recent arterial cannulation (i.e., less than 30 days prior to study date)
* Six or more arterial cannulations of each (right & left) radial artery
* History of clinically significant complications from previous arterial cannulation
* Current use of blood thinners: prescription or daily aspirin use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Up to 20 subjects recruited from the Clinical Laboratory subject data base.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pulse oximetry measurements of saturation from the test device will be compared to CO-Oximetry measurements of arterial oxygen saturation to demonstrate that the test sensor meets the oxygen saturation accuracy specifications for SpO2. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Heyer, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Boulder Clinical Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No